CLINICAL TRIAL: NCT05404971
Title: Effects of Joint Integrity Exercises Verses Mirror Therapy on Proprioception and Functional Rehabilitation of Upper Limb in Hemineglect Stroke Survivors
Brief Title: Effects of Joint Integrity Exercises Verses Mirror Therapy in Hemineglect Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/21/0210 Faiza Tabassam
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Stroke
Keywords: Joint integrity ,Proprioception, Mirror therapy, Hemineglect
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Joint integrity exercises (Experimental): Tactile stimulation with the various textures will be applied to the patients with three strokes followed by 3 sec rest period.
  Kinaesthetic stimulations will be given to the patients to increase proprioception proprioception in neglected limb in sitting position, the limb on the affected side of the body is supported and moved by the examiner in various directions but movement is only at one joint at a time. Stereognosis by placing the object in the patient's hand for a maximum 30 seconds with close eyes. Identification is by naming, description or by pair matching with an identical set.
  Interventions: Other: Joint integrity exercises
- Mirror therapy (Active Comparator): A 5 cm × 35 cm mirror will be placed vertically between the upper limbs on the table, with the reflecting surface facing the uninjured limb. Patients will be asked to observe the motion of the upper limb on the uninjured side and imagine that the limb on the affected side was in motion, imagine the motion of the affected limb the same as that observed on the uninjured side, and complete 6 movements including shoulder joint forward flexion, elbow joint flexion and extension, forearm forward and backward rotation, wrist joint flexion and extension, finger extension and grasping, and thumb abduction. The participants will be asked to perform each movement for 5 min and try to reach the maximum range of motion of the joints. Training will be completed for 30 min per day) Session will be 3 days per week. Per day session will be for 30 minutes.
  Interventions: Other: Mirror therapy

INTERVENTIONS:
Other: Joint integrity exercises — patients with three strokes followed by 3 sec rest period. Kinaesthetic stimulations will be given to the patients to increase proprioception proprioception in neglected limb in sitting position, the limb on the affected side of the body is supported and moved by the examiner in various directions but movement is only at one joint at a time. Stereognosis by placing the object in the patient's hand for a maximum 30 seconds with close eyes. Identification is by naming, description or by pair matching with an identical set.
  Arms: Joint integrity exercises
Other: Mirror therapy — A 5 cm × 35 cm mirror will be placed vertically between the upper limbs on the table, with the reflecting surface facing the uninjured limb. Patients will be asked to observe the motion of the upper limb on the uninjured side and imagine that the limb on the affected side was in motion, imagine the motion of the affected limb the same as that observed on the uninjured side, and complete 6 movements including shoulder joint forward flexion, elbow joint flexion and extension, forearm forward and backward rotation, wrist joint flexion and extension, finger extension and grasping, and thumb abduction. The participants will be asked to perform each movement for 5 min and try to reach the maximum range of motion of the joints. Training will be completed for 30 min per day) Session will be 3 days per week. Per day session will be for 30 minutes.
  Arms: Mirror therapy

SUMMARY:
The aim of this study is to compare the effects of joint integrity exercises and mirror therapy to evaluate that which intervention is more effective to improve proprioception and motor function of upper limb in hemineglect stroke survivors. This will be randomized clinical triall study. Data will be collected from Lahore General Hospital by using non-probability convenient sampling technique. Patients will be divided into two groups, (Group A and Group B). Group A will include patients that will be treated with joint integrity exercises of upper limb by applying tactile stimulation, kinaesthetic stimulation and stereognosis. and Group B will include those patients which will be treated with mirror therapy of upper limb. Session will be 3 days per week. Data will be collected pre (baseline=0 week) and post intervention (after 6 weeks) from two groups using Nottingham sensory assessment, Fugl Mayer Assessment and Motor assessment scale. SPSS for windows software, version 25 will be used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* Hemi neglect stroke patients after performing line bisection test
* Patients having Mini mental State Examination score above 24
* Patients having Catherine Bergego scale score above 27
* Patients having minimum MIQ-3 score 6 or above
* Sub-acute phase (2 Months) following stroke

Exclusion Criteria:

* Patients with neurological conditions other than stroke including Parkinson's, Alzheimer and Multiple sclerosis

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity Assessment | 4 weeks
  The Fugl-Meyer Upper Extremity (FMUE) Scale is a widely used and highly recommended stroke-specific, performance-based measure of impairment. It is used for assessment of motor function of upper extremity. The FMUE Scale comprises 33 items, each item scored on 3 point ordinal scale of 0 to 2, where 0 = cannot perform, 1 = performs partially and 2 = performs fully. Total score for motor function is 66. Reading will be at Baseline and after 4 weeks
Nottingham sensory assessment | 4 weeks
  NSA is used in clinical trials in stroke patients to test effectiveness of different interventions. It is used for sensory examination of tactile sensation, kinesthesia and stereognosis. Tactile scoring is 0-2, where 0 = absent, 1 = impaired and 2 = normal. Stereognosis scoring is 0-2, where 0 = absent, 1 = impaired and 2 = normal. Kinesthesia scoring 0-3, where 0 = absent, 1 = appreciation of movement taking place, 2 = direction of movement sense and 3 = joint position sense.
  Reading will be at Baseline and after 4 weeks
Motor assessment scale | 4 weeks
  This scale is designed to assess the return of function following a stroke or other neurological impairment. The test looks at a patient's ability to move with low tone or in a synergistic pattern and finally move actively out of that pattern into normal movement. It consists of 9 sections. The higher the score, the higher functioning the patient has on the affected side. High Score = 54 and Low Score = 0.
  Reading will be at Baseline and after 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tehreem Mukhtar, MS, Principal Investigator — Riphah International University
Locations (1):
- Lahore General Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Veerbeek JM, van Wegen E, van Peppen R, van der Wees PJ, Hendriks E, Rietberg M, Kwakkel G. What is the evidence for physical therapy poststroke? A systematic review and meta-analysis. PLoS One. 2014 Feb 4;9(2):e87987. doi: 10.1371/journal.pone.0087987. eCollection 2014. PMID 24505342
- [Background] Campbell BCV, De Silva DA, Macleod MR, Coutts SB, Schwamm LH, Davis SM, Donnan GA. Ischaemic stroke. Nat Rev Dis Primers. 2019 Oct 10;5(1):70. doi: 10.1038/s41572-019-0118-8. PMID 31601801
- [Background] Harrison DH, DeVore BB, Campbell RW, Harrison PK. Hallucinations and hemispatial neglect following right middle cerebral artery cerebrovascular accident: Left gaze bias with left sensory hemineglect syndrome. 2017